CLINICAL TRIAL: NCT06921668
Title: Perioperative Dynamics of Energy Expenditure in Lewis-Santy Oesophagectomy Patients
Brief Title: Perioperative Dynamics of Energy Expenditure in Oesophagectomy Patients
Acronym: OESOCAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0271/OB; IDRCB : 2023-A02724-41 (Other: ANSM)
Record Dates: First submitted 2025-03-19; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Oesophagectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Carcinological oesophageal resection surgery is one of the so-called major digestive surgeries, i.e. involving a high perioperative risk (morbidity and mortality) in patients who are malnourished or at high risk of malnutrition.

Nutritional therapy for these patients is an important part of overall perioperative management. Lewis-Santy oesophageal surgery requires a thoracic approach (thoracotomy or thoracoscopy) and an abdominal approach (laparotomy or laparoscopy).

Resumption of oral feeding is contraindicated in the immediate postoperative period. The use of a feeding jejunostomy is not systematic. The methods used to manage artificial nutritional support vary between centres, but the foreseeable duration of fasting and/or intake of less than 50% of nutritional requirements is always greater than 5 days.

At present, total energy requirements are calculated using formulae that take into account the patient's inflammatory state (stable, unstable or stabilised patient), theoretical ideal weight and previous nutritional status, in order to come as close as possible to actual energy expenditure, and are the subject of perioperative nutrition protocols specific to each centre. Indirect calorimetry makes it possible to reliably measure energy expenditure during the perioperative period.

The OESOCAL study continues this line of reasoning. It assumes that energy expenditure may vary according to the surgical approach, and that indirect calorimetry can be used to optimise nutritional support in order to avoid over- or under-nutrition, which may be responsible for an increase in infectious complications.

DETAILED DESCRIPTION:
The results of this study should enable current nutrition protocols to evolve and nutritional support to be incorporated into a more global project of individualised perioperative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted for scheduled digestive surgery for Lewis Santy oesophagectomy whose care pathway includes a stay in an intensive care unit or continuing care unit.
* Member or beneficiary of a social protection scheme
* Patient who has read and understood the information letter and does not object to taking part in the study.

Exclusion Criteria:

* Contraindication to indirect calorimetry (oxygen therapy, etc.)
* Refusal to take part in the study
* No social security affiliation
* Patient is a minor
* Patient under legal protection (guardianship)
* Pregnant women
* Oesophagectomy with cervical approach (3-way oesophagectomy)
* Participation in an interventional research protocol likely to have an effect on perioperative nutritional status or surgical technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patient admitted for digestive surgery for Lewis Santy oesophagectomy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Determining perioperative dynamics of energy expenditure | Perioperative resting energy expenditure: preoperatively on Day-21/Day-15 or Day-1 of the operation and postoperatively on Day2-Day4 and Day6-Day8
  Describe the perioperative dynamics of energy expenditure in patients undergoing Lewis-Santy carcinological oesophagectomy as a function of surgical technique by indirect calorimetry (assessing resting energy expenditure ).

SECONDARY OUTCOMES:
Total nutritional intake (vitamin intake) | pre-operatively on Day-21/Day-15 or Day-1 of the operation and post-operatively on Day2-Day4
  Assessing patients' total nutritional intake in the perioperative period
Total nutritional intake (parenteral/enteral nutrition) | pre-operatively on Day-21/Day-15 or Day-1 of the operation and post-operatively on Day2-Day4
  Post-operative nutritional support: parenteral/enteral nutrition intake
Total nutritional intake (Trace elements) | pre-operatively on Day-21/Day-15 or Day-1 of the operation and post-operatively on Day2-Day4
  Post-operative nutritional support: trace elements intake
Comparison of calorie targets set with data measured by indirect calorimetry | Perioperative resting energy expenditure: preoperatively on Day-21/Day-15 or Day-1 of the operation and postoperatively on Day2-Day4 and Day6-Day8
  Comparison of calorie targets set by the postoperative artificial nutrition protocol with data measured by indirect calorimetry
Post-operative complications | at 6 and 12 months
  Postoperative morbidity and mortality, surgical complications evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Emilie EO OCCHIALI, Doctor, Study Chair — Surgical Intensive Care Unit, UH of Rouen
Locations (4):
- France (4):
  - Service d'Anesthésie-Réanimation, Amiens
  - Department of Anaesthesia and Intensive Care, Brest
  - Surgical Intensive Care Department, Rouen
  - Department of Anaesthesia, Intensive Care and Perioperative Medicine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.